CLINICAL TRIAL: NCT05464875
Title: A Multicenter Study of Avapritinib Efficacy and Safety of Metastatic or Unresectable Gastrointestinal Stromal Tumors
Status: Recruiting | Type: Observational
Sponsor: Xinhua Zhang, MD (Other)
Collaborators: Peking University Cancer Hospital & Institute (Other); Fudan University (Other); Peking University People's Hospital (Other); Chinese PLA General Hospital (Other); Xiangya Hospital of Central South University (Other); Peking University Shenzhen Hospital (Other); Nanfang Hospital, Southern Medical University (Other); West China Hospital (Other); Jiangsu Cancer Institute & Hospital (Other); Shanghai Zhongshan Hospital (Other); Sun Yat-sen University (Other); Xijing Hospital (Other); Shengjing Hospital (Other); Shanghai Jiao Tong University School of Medicine (Other); Liaoning Cancer Hospital & Institute (Other); Sixth Affiliated Hospital, Sun Yat-sen University (Other); Fujian Medical University Union Hospital (Other); Cancer Hospital of Guangxi Medical University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); First Affiliated Hospital of Chongqing Medical University (Other); Chongqing University Cancer Hospital (Other)
Responsible Party: Sponsor-Investigator, Xinhua Zhang, MD, First Affiliated Hospital, Sun Yat-Sen University, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Other Study IDs: No.[2022]106
Record Dates: First submitted 2022-07-09; First posted 2022-07-19 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Gastrointestinal Stromal Tumors; Unresectable Solid Tumor; Recurrent Metastatic Malignant Neoplasm
Keywords: Avapritinib; Genetic testing
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a prospective, multicenter, observational real-world study to explore the therapy patterns and clinical outcomes of Avapritinib in patients with metastatic or unresectable gastrointestinal stromal tumors.

DETAILED DESCRIPTION:
INTRODUCTION AND RATIONALE Gastrointestinal stromal tumors (GIST) are thought to develop from the interstitial cells of Cajal or their stem cell precursors. They are the most common mesenchymal tumors occurring in the gastrointestinal (GI) tract. The annual incidence of GIST is about 1/100,000 ~ 2/100,000 globally. Biological behavior can range from benign to malignant, and immunohistochemical staining is usually positive for CDs 117 and DOG-1, showing Cajal cell differentiation. Eighty-five percent of GISTs is caused by activating mutations in the receptor tyrosine kinase KIT or platelet-derived growth factor receptor alpha (PDGFRA) gene. Targeted therapy for KIT and PDGFRA alters metastatic or unresectable GISTs without effective drug therapy, allowing tumor control and significantly prolonging patient survival. Imatinib, a first-line drug, has been shown to control in 80% of patients, whereas 50% of patients develop tumor progression after twenty-four months of treatment, with an estimated ten-year progression-free survival (PFS) rate of approximately 9 %. The most significant cause of progression was secondary mutations in the ATP binding domain or activation ring of KIT results in resistance to imatinib. Sunitinib, the second-line standard of care, and regorafenib, the third-line standard of care, inhibit some of the secondary mutations, with median PFSs of about 5.6 months for sunitinib and 4.8 months for regorafenib. However, imatinib and other targeted drugs that have been approved for the treatment of GISTs are naturally resistant to the activated ring exon 18 D842V mutation of PDGFRA, which accounts for 5 %-6 %[10% of the primary mutations in GISTs. Avapritinib was approved for marketing in January 2020 for the treatment of PDGFRA D842V mutant GISTs, thus making this type of GISTs medically acceptable.

Avapritinib is a type I tyrosine kinase inhibitor (TKI) that has significant inhibitory effects on KIT or PDGFRA in activated configurations, such as mutations in the KIT or PDGFRA activated loop. Preclinical studies have found broad-spectrum inhibition of KIT or PDGFRA, including mutations in exons 11,17,18 of KIT, and mutations in exon 18 of PDGFRA, with a 24 hr, concentration-dependent inhibitory effect. Weak affinity for wild-type KIT and PDGFRA, PDGFRB, CSF1R, and FLT3. In the Phase 1 clinical study in patients with metastatic or unresectable PDGFRA D842V-mutated GISTs, the objective response rate (ORR) for avapritinib was 91%, with a complete response rate of 13%, a median duration of efficacy (DOR) of 27.6 m (95% CI 17.6-N%), and a median PFS of 34 m (95% CI 22.9-N%) estimated to be 61% at 36months. The daily 30-600 mg of Avapritinib showed an initial anti-tumor effect, but the time to effect at the high dose was significantly shorter than at the low dose. Both the US and the European Medicines Agency (FDA and EMA) have approved the use of Avapritinib in GISTs with PDGFRA exon 18 mutations due to its significant therapeutic effect on PDGFRA D842V mutations. In patients with KIT or non-D842V PDGFRA mutations treated more than three lines, the ORRs of atorvastatin were 17%, all were partial responses (PRs), the median DORs were 10.2 m (95% CI 7.% -10.2), the clinical benefit rate (CBRs) was 38%, the median PFSs were 3.7 m (95% CI 2.% -4.6), the median OSs were 11.6 m (95% CI 9.% -12.6), and there was no difference in efficacy between the 300 mg and 400 mg daily dose groups. The above studies showed that Avapritinib was effective in the treatment of PDGFRA D842V mutant GISTs, and some patients with KIT or non-D842V PDGFRA mutations were able to obtain tumor control from the treatment of Avapritinib, with a dose effect on the anti-tumor efficacy, but no significant difference in the high dose 300 mg or 400 mg efficacy.

With respect to the safety of avapritinib, patients with >99% reported at least one adverse event (Adverse events, AEs), with common AEs including nausea (59%), fatigue (50%), periorbital edema (42%), anemia (39%), diarrhea (36%), and vomiting (33%). The incidence of grade ≥3 AEs was 72% and higher in the 400 mg dose group than in the 300 mg dose group, 84% and 73%, respectively. Common AEs included anemia (30%), fatigue (8%), abdominal pain (6%) and hypophosphatemia (6%). The incidence and severity of AEs in elderly patients (≥65 y) was slightly higher than that in younger patients. The incidence of treatment-related adverse events leading to discontinuation of Avapritinib was 11.2%, the most common were cognitive effects (4.1%), intracranial hemorrhage (1.2%), fatigue (<1%), and vomiting (<1%), which were higher in the 400 mg group than in the 300 mg group. The incidence of downtitration of Avapritinib was (32%), and the incidence of AEs of each grade and grade ≥3 was significantly lower after downtitration than before downtitration.

Preclinical studies with avapritinib suggest that the drug can penetrate the blood-brain barrier with a brain-to-plasma concentration ratio of 0.7 -1.0 3, leading to edema of the choroid plexus in dogs and intracranial hemorrhage at high doses. Therefore, central nervous system AEs, including cognitive effects and intracranial haemorrhage [14], are of particular interest in clinical studies. In the Phase I/II clinical study of Avapritinib (Navigator), the incidence of cognitive effects in patients receiving Avapritinib was 42% (104/250) and 40% in the 300 mg group, which was lower than that in the 400 mg dose group (50%). Memory impairment was the most common manifestation of cognitive effects, with an incidence of 27% in the 300 mg group and 40% in the 400 mg group, with a higher incidence in elderly patients (age ≥65 y). The cognitive effects were mostly Grade 1-2 in the Avapritinib 300 mg group and 7.5% in the Avapritinib 300 mg group. The cognitive effects were improved in most patients by discontinuation or dose adjustment, with a median adjusted dose of 233 mg. The incidence of intracranial hemorrhage was 2.4% in the Avapritinib 300 mg dose group, one case of grade 1 subdural hematoma, three cases of grade 1, 2 and 4 intracranial hemorrhage, and one case of grade 3 intracranial hemorrhage. Intracranial hemorrhage was improved by discontinuation or dose adjustment, and no patient died due to intracranial hemorrhage. Median PFSs were 11.4 m (95 %CI 8.% -20.3) in dose-reduced patients and 7.2 m (95 %CI 5.% -24.0) in dose-unadjusted patients, with similar trends for both non-D842V 4 + line therapy and D842V mutations. These studies indicate that the overall safety of Avapritinib is adequate, but special attention needs to be paid to central nervous system AEs, including cognitive abnormalities and cerebral haemorrhage, which have a dose effect, the incidence of high-dose cognitive abnormalities of Avapritinib is higher, the incidence of high-dose cognitive abnormalities of Avapritinib is higher after dose reduction, whether D842V mutations or non-D842V mutations, dose adjustment does not affect survival, and PFSs are longer in appropriately reduced-dose patients.

Avapritinib is a small molecule oral TKI with a dose-proportional increase in Cmax and AUC over the 30-400 mg qd range with a mean accumulation rate of 2. -8.9 2 after repeat dosing. Protein binding was 98.8%, mainly metabolized by CYP3A in vivo, 70% excreted in feces, major metabolite, and plasma elimination half-life was 32-57 h. Pharmacokinetic inter-individual differences were large, with in vivo exposure varying up to 8-10-fold in the 300 mg qd dose group. Approximately 50% or more of the patients who started 300 mg qd had high drug exposures, and the incidence of cognitive abnormalities was associated with cumulative exposure to Avapritinib, i.e., there were large individual pharmacokinetic differences, with a tendency to increase the incidence of Grade III or IV AEs as patients' in vivo concentrations of Avapritinib increased. However, there are no lowest effective exposures and highest toxic exposures leading to central nervous AEs in the benefit populations of atorvastatin for the treatment of PDGFRA D842V mutations and PDGFRA mutations with KIT or non-D842V.

Therefore, it is necessary to conduct a multicenter observational study on the pharmacokinetics, efficacy, and safety of Avapritinib in patients with metastatic or unresectable GIST, to explore the influencing factors on the pharmacokinetics of Avapritinib, to identify the treatment window of Avapritinib, so that the dose can be adjusted according to the in vivo exposure of Avapritinib, to reduce the risk or severity of AEs, to improve the treatment effect, and to conduct individualized administration.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are aged ≥ 18 years.
* Gastrointestinal stromal tumors confirmed by histopathological examination, and CD- and/or DOG-1-positive by immunohistochemistry.
* Presence of mRECIST v1.1-compliant lesions with at least one measurable lesion (non-lymphadenopathy ≥1.0 cm or ≥2-fold scan slice thickness).
* Treatment with Avapritinib.
* Patients with an Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 to 2 at screening.
* Patient informed consent and signed written consent form.
* The patient was compliant and voluntarily scheduled for follow-up, treatment, laboratory tests, and other study procedures.

Exclusion Criteria:

* KIT or PDGFRA wild type.
* Failure to complete continuous atorvastatin for at least 15 days due to intolerability or disease progression.
* Other serious acute or chronic physical or mental problems, or laboratory abnormalities, may increase the risk associated with participation in the study or use of drugs, or interfere with the judgment of the study results and, in the judgment of the investigator, are not considered appropriate for participation in the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 74 patients with metastatic or unresectable advanced gastrointestinal stromal tumors from tier-3 hospitals who meet the criteria will be enrolled in the study.
Sampling Method: Probability Sample
Enrollment: 74 (Estimated)
Dates: Start 2022-07-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 2 years
  To evaluate objective response rate (ORR,CR+PR) determined by radiology assessment per mRECIST(Response Evaluation Criteriain Solid Tumours), version 1.1 in patients with Metastatic or Unresectable Gastrointestinal Stromal Tumors.Complete response is the disappearance of all lesions with nodes measuring < 10 mm and normal tumour markers.A decrease in the sum of target disease of ≥ 30% represents partial response.
Clinical Benefit Rate | 2 years
  To evaluate clinical benefit rate(CBR,CR+PR+>16 weeks continuation SD) determined by radiology assessment per mRECIST, version 1.1 in patients with Metastatic or Unresectable Gastrointestinal Stromal Tumors.Complete response is the disappearance of all lesions with nodes measuring < 10 mm and normal tumour markers.A decrease in the sum of target disease of ≥ 30% represents partial response.Stable disease lies between partial response and progressive disease.
Duration Of Response | 2 years
  To evaluate duration of response (DOR) determined by radiology assessment per mRECIST, version 1.1 in patients with Metastatic or Unresectable Gastrointestinal Stromal Tumors.Complete response is the disappearance of all lesions with nodes measuring < 10 mm and normal tumour markers.A decrease in the sum of target disease of ≥ 30% represents partial response.Stable disease lies between partial response and progressive disease.If a lesion reappears after disappearing in a patient with complete response, progressive disease is declared. However, if such a lesion behaves in this manner in a patient with stable disease or partial response, it is the change in sum of target disease that defines the response or progression.

SECONDARY OUTCOMES:
Progression-free survival | 2 years
  To evaluate PFS determined by radiology assessment per mRECIST, version 1.1 in patients with Metastatic or Unresectable Gastrointestinal Stromal Tumors.Complete response is the disappearance of all lesions with nodes measuring < 10 mm and normal tumour markers.A decrease in the sum of target disease of ≥ 30% represents partial response.Stable disease lies between partial response and progressive disease.If a lesion reappears after disappearing in a patient with complete response, progressive disease is declared. However, if such a lesion behaves in this manner in a patient with stable disease or partial response, it is the change in sum of target disease that defines the response or progression.
overall survival | 2 years
  To evaluate OS determined in patients with Metastatic or Unresectable Gastrointestinal Stromal Tumors.Complete response is the disappearance of all lesions with nodes measuring < 10 mm and normal tumour markers.A decrease in the sum of target disease of ≥ 30% represents partial response.Stable disease lies between partial response and progressive disease.If a lesion reappears after disappearing in a patient with complete response, progressive disease is declared. However, if such a lesion behaves in this manner in a patient with stable disease or partial response, it is the change in sum of target disease that defines the response or progression.
Treatment-emergent adverse events | 2 years
  To evaluate treatment-emergent adverse events determined in patients with Metastatic or Unresectable Gastrointestinal Stromal Tumors.
adverse events of special interest | 2 years
  To evaluate adverse events of special interest determined in patients with Metastatic or Unresectable Gastrointestinal Stromal Tumors.
serious adverse events | 2 years
  To evaluate serious adverse events determined in patients with Metastatic or Unresectable Gastrointestinal Stromal Tumors.
t1/2 | 2 years
  To evaluate t1/2 determined in patients with Metastatic or Unresectable Gastrointestinal Stromal Tumors.t1/2:The half-life of a drug is the time it takes to metabolize half of a drug.
Cmin(minimum concentration) | 2 years
  To evaluate minimum concentration determined in patients with Metastatic or Unresectable Gastrointestinal Stromal Tumors.
Cmax(Peak Concentration) | 2 years
  To evaluate Peak Concentration determined in patients with Metastatic or Unresectable Gastrointestinal Stromal Tumors.
Css,avg（Mean blood drug concentration） | 2 years
  To evaluate Mean blood drug concentration determined in patients with Metastatic or Unresectable Gastrointestinal Stromal Tumors.
Tmax（peak time） | 2 years
  To evaluate peak time determined in patients with Metastatic or Unresectable Gastrointestinal Stromal Tumors.
AUC（area under the curve） | 2 years
  To evaluate area under the curve determined in patients with Metastatic or Unresectable Gastrointestinal Stromal Tumors.
CL（clearance rate） | 2 years
  To evaluate clearance rate determined in patients with Metastatic or Unresectable Gastrointestinal Stromal Tumors.
Vd（volume of distribution） | 2 years
  To evaluate volume of distribution determined in patients with Metastatic or Unresectable Gastrointestinal Stromal Tumors.

OTHER OUTCOMES:
resistance gene mutation status | 2 years
  Analysis of resistance gene mutation status in the treated population verse before the treatment by gene testing.
Assessment of dose effect of antineoplastic agents | 2 years
  The clinical effects of anti-tumor drugs in the treated population were assessed by monitoring according to the pharmacokinetic indicators mentioned above.

CONTACTS AND LOCATIONS:
Overall Officials: Xinhua Zhang, PhD, Principal Investigator — First affiliated hosptial,Sun Yat-sen university
Locations (1):
- The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fletcher CD, Berman JJ, Corless C, Gorstein F, Lasota J, Longley BJ, Miettinen M, O'Leary TJ, Remotti H, Rubin BP, Shmookler B, Sobin LH, Weiss SW. Diagnosis of gastrointestinal stromal tumors: A consensus approach. Hum Pathol. 2002 May;33(5):459-65. doi: 10.1053/hupa.2002.123545. PMID 12094370
- [Background] von Mehren M, Joensuu H. Gastrointestinal Stromal Tumors. J Clin Oncol. 2018 Jan 10;36(2):136-143. doi: 10.1200/JCO.2017.74.9705. Epub 2017 Dec 8. PMID 29220298
- [Background] China Society of Clinical Oncology Gastrointestinal Stromal Tumors Expert Committee. Chinese Consensus on Diagnosis and Treatment of Gastrointestinal Stromal Tumors (2017 Edition). Electronic Journal of Comprehensive Cancer Therapy. 2018;4(1): 31-42.
- [Background] Ducimetiere F, Lurkin A, Ranchere-Vince D, Decouvelaere AV, Peoc'h M, Istier L, Chalabreysse P, Muller C, Alberti L, Bringuier PP, Scoazec JY, Schott AM, Bergeron C, Cellier D, Blay JY, Ray-Coquard I. Incidence of sarcoma histotypes and molecular subtypes in a prospective epidemiological study with central pathology review and molecular testing. PLoS One. 2011;6(8):e20294. doi: 10.1371/journal.pone.0020294. Epub 2011 Aug 3. PMID 21826194
- [Background] Heinrich MC, Corless CL, Demetri GD, Blanke CD, von Mehren M, Joensuu H, McGreevey LS, Chen CJ, Van den Abbeele AD, Druker BJ, Kiese B, Eisenberg B, Roberts PJ, Singer S, Fletcher CD, Silberman S, Dimitrijevic S, Fletcher JA. Kinase mutations and imatinib response in patients with metastatic gastrointestinal stromal tumor. J Clin Oncol. 2003 Dec 1;21(23):4342-9. doi: 10.1200/JCO.2003.04.190. PMID 14645423
- [Background] Casali PG, Zalcberg J, Le Cesne A, Reichardt P, Blay JY, Lindner LH, Judson IR, Schoffski P, Leyvraz S, Italiano A, Grunwald V, Pousa AL, Kotasek D, Sleijfer S, Kerst JM, Rutkowski P, Fumagalli E, Hogendoorn P, Litiere S, Marreaud S, van der Graaf W, Gronchi A, Verweij J; European Organisation for Research and Treatment of Cancer Soft Tissue and Bone Sarcoma Group, Italian Sarcoma Group, and Australasian Gastrointestinal Trials Group. Ten-Year Progression-Free and Overall Survival in Patients With Unresectable or Metastatic GI Stromal Tumors: Long-Term Analysis of the European Organisation for Research and Treatment of Cancer, Italian Sarcoma Group, and Australasian Gastrointestinal Trials Group Intergroup Phase III Randomized Trial on Imatinib at Two Dose Levels. J Clin Oncol. 2017 May 20;35(15):1713-1720. doi: 10.1200/JCO.2016.71.0228. Epub 2017 Mar 31. PMID 28362562
- [Background] Wardelmann E, Merkelbach-Bruse S, Pauls K, Thomas N, Schildhaus HU, Heinicke T, Speidel N, Pietsch T, Buettner R, Pink D, Reichardt P, Hohenberger P. Polyclonal evolution of multiple secondary KIT mutations in gastrointestinal stromal tumors under treatment with imatinib mesylate. Clin Cancer Res. 2006 Mar 15;12(6):1743-9. doi: 10.1158/1078-0432.CCR-05-1211. PMID 16551858
- [Background] Demetri GD, van Oosterom AT, Garrett CR, Blackstein ME, Shah MH, Verweij J, McArthur G, Judson IR, Heinrich MC, Morgan JA, Desai J, Fletcher CD, George S, Bello CL, Huang X, Baum CM, Casali PG. Efficacy and safety of sunitinib in patients with advanced gastrointestinal stromal tumour after failure of imatinib: a randomised controlled trial. Lancet. 2006 Oct 14;368(9544):1329-38. doi: 10.1016/S0140-6736(06)69446-4. PMID 17046465
- [Background] Demetri GD, Reichardt P, Kang YK, Blay JY, Rutkowski P, Gelderblom H, Hohenberger P, Leahy M, von Mehren M, Joensuu H, Badalamenti G, Blackstein M, Le Cesne A, Schoffski P, Maki RG, Bauer S, Nguyen BB, Xu J, Nishida T, Chung J, Kappeler C, Kuss I, Laurent D, Casali PG; GRID study investigators. Efficacy and safety of regorafenib for advanced gastrointestinal stromal tumours after failure of imatinib and sunitinib (GRID): an international, multicentre, randomised, placebo-controlled, phase 3 trial. Lancet. 2013 Jan 26;381(9863):295-302. doi: 10.1016/S0140-6736(12)61857-1. Epub 2012 Nov 22. PMID 23177515
- [Background] Corless CL, Schroeder A, Griffith D, Town A, McGreevey L, Harrell P, Shiraga S, Bainbridge T, Morich J, Heinrich MC. PDGFRA mutations in gastrointestinal stromal tumors: frequency, spectrum and in vitro sensitivity to imatinib. J Clin Oncol. 2005 Aug 10;23(23):5357-64. doi: 10.1200/JCO.2005.14.068. Epub 2005 May 31. PMID 15928335
- [Background] Klug LR, Kent JD, Heinrich MC. Structural and clinical consequences of activation loop mutations in class III receptor tyrosine kinases. Pharmacol Ther. 2018 Nov;191:123-134. doi: 10.1016/j.pharmthera.2018.06.016. Epub 2018 Jun 30. PMID 29964125
- [Background] Evans EK, Gardino AK, Kim JL, Hodous BL, Shutes A, Davis A, Zhu XJ, Schmidt-Kittler O, Wilson D, Wilson K, DiPietro L, Zhang Y, Brooijmans N, LaBranche TP, Wozniak A, Gebreyohannes YK, Schoffski P, Heinrich MC, DeAngelo DJ, Miller S, Wolf B, Kohl N, Guzi T, Lydon N, Boral A, Lengauer C. A precision therapy against cancers driven by KIT/PDGFRA mutations. Sci Transl Med. 2017 Nov 1;9(414):eaao1690. doi: 10.1126/scitranslmed.aao1690. PMID 29093181
- [Background] Gebreyohannes YK, Wozniak A, Zhai ME, Wellens J, Cornillie J, Vanleeuw U, Evans E, Gardino AK, Lengauer C, Debiec-Rychter M, Sciot R, Schoffski P. Robust Activity of Avapritinib, Potent and Highly Selective Inhibitor of Mutated KIT, in Patient-derived Xenograft Models of Gastrointestinal Stromal Tumors. Clin Cancer Res. 2019 Jan 15;25(2):609-618. doi: 10.1158/1078-0432.CCR-18-1858. Epub 2018 Oct 1. PMID 30274985
- [Background] Heinrich MC, Jones RL, von Mehren M, Schoffski P, Serrano C, Kang YK, Cassier PA, Mir O, Eskens F, Tap WD, Rutkowski P, Chawla SP, Trent J, Tugnait M, Evans EK, Lauz T, Zhou T, Roche M, Wolf BB, Bauer S, George S. Avapritinib in advanced PDGFRA D842V-mutant gastrointestinal stromal tumour (NAVIGATOR): a multicentre, open-label, phase 1 trial. Lancet Oncol. 2020 Jul;21(7):935-946. doi: 10.1016/S1470-2045(20)30269-2. PMID 32615108
- [Background] Jones RL, Serrano C, von Mehren M, George S, Heinrich MC, Kang YK, Schoffski P, Cassier PA, Mir O, Chawla SP, Eskens FALM, Rutkowski P, Tap WD, Zhou T, Roche M, Bauer S. Avapritinib in unresectable or metastatic PDGFRA D842V-mutant gastrointestinal stromal tumours: Long-term efficacy and safety data from the NAVIGATOR phase I trial. Eur J Cancer. 2021 Mar;145:132-142. doi: 10.1016/j.ejca.2020.12.008. Epub 2021 Jan 16. PMID 33465704
- [Background] George S, Jones RL, Bauer S, Kang YK, Schoffski P, Eskens F, Mir O, Cassier PA, Serrano C, Tap WD, Trent J, Rutkowski P, Patel S, Chawla SP, Meiri E, Gordon M, Zhou T, Roche M, Heinrich MC, von Mehren M. Avapritinib in Patients With Advanced Gastrointestinal Stromal Tumors Following at Least Three Prior Lines of Therapy. Oncologist. 2021 Apr;26(4):e639-e649. doi: 10.1002/onco.13674. Epub 2021 Feb 1. PMID 33453089
- [Background] Joseph CP, Abaricia SN, Angelis MA, Polson K, Jones RL, Kang YK, Riedel RF, Schoffski P, Serrano C, Trent J, Tetzlaff ED, Si TD, Zhou T, Doyle A, Bauer S, Roche M, Havnaer T. Optimal Avapritinib Treatment Strategies for Patients with Metastatic or Unresectable Gastrointestinal Stromal Tumors. Oncologist. 2021 Apr;26(4):e622-e631. doi: 10.1002/onco.13632. Epub 2021 Jan 5. PMID 33301227
- [Background] Trullas-Jimeno A, Delgado J, Garcia-Ochoa B, Wang I, Sancho-Lopez A, Payares-Herrera C, Dalhus ML, Strom BO, Egeland EJ, Enzmann H, Pignatti F. The EMA assessment of avapritinib in the treatment of gastrointestinal stromal tumours harbouring the PDGFRA D842V mutation. ESMO Open. 2021 Jun;6(3):100159. doi: 10.1016/j.esmoop.2021.100159. Epub 2021 May 20. PMID 34023541
- [Background] Joseph CP, Abaricia SN, Angelis MA et al. Avapritinib for the treatment of GIST: Analysis of efficacy, safety, and patient management strategies at the recommended phase 2 dose. Presented at: Connective Tissue Oncology Society Annual Meeting; 2019; Tokyo, Japan.